CLINICAL TRIAL: NCT04176861
Title: Home-based Brainwave Entrainment Technology (hBET) for Management of Chronic Pain and Sleep Disturbance: A Feasibility Study.
Brief Title: hBET for Pain and Sleep Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Leeds (Other)
Responsible Party: Principal Investigator, Stephen Halpin, Visiting Clinical Research Fellow, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NHS001542
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pain, Chronic; Sleep Disturbance
Keywords: audio-visual stimulation; brainwave entrainment
MeSH Terms: conditions — Chronic Pain; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Home based intervention (Experimental): Participants using hBET technology at home (all participants).
  Interventions: Device: home-based Brainwave Entrainment Technology

INTERVENTIONS:
Device: home-based Brainwave Entrainment Technology — Smartphone app-based brainwave entrainment programme using audio stimulation via binaural beats or visual stimulation via flickering lights

SUMMARY:
Long-term pain affects one-third of the United Kingdom population and can be very disabling. People experiencing long-term pain often suffer from disturbed sleep because of their pain symptoms, and disturbed sleep can then make their pain symptoms worse. Managing long-term pain is also very costly to the National Health Service. The most common treatment is prescribed medicines, but these do not always work and can have serious side-effects for some patients.

The investigators have been developing an alternative approach for treating long-term pain. This approach uses simple non-invasive tools to promote some kinds of brain activity over others. It involves patients using headphones to listen to some specific sounds, or a headset with lights flashing at particular frequencies. The studies undertaken so far seem to show that doing this can change how the brain responds to pain. It potentially offers an inexpensive yet effective way of reducing pain and improving sleep for patients with long-term pain. There are a few small studies that support this approach and more work is needed. The next step is to find out whether these tools can be reliably used in home settings, how people feel about using this approach, and to gather information to design a larger trial of this technology.

Therefore the aim of this study is to test the suitability and acceptability of these home-based tools with individuals with long-term pain. Up to 30 participants with long-term pain and pain-related sleep disturbance will use the tools for at least 20 minutes at bed time every day for 4 weeks. The investigators will interview them to ask about their experiences of using the tools, and their feedback and suggestions on how the approach should be developed. The investigators will measure changes in the nature of participants' pain, sleep, fatigue and mood.

These findings will inform the planning and design of a future much larger study to test this technology. The investigators will make sure that findings from this study are shared widely within the National Health Service and beyond among patient groups, professionals, charities, specialist centres and commissioners.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-cancer pain (recurring pain ≥ 3 months duration)
* Having nocturnal pain (NRS 0-10 worst pain ≥ 4)
* Self-reported sleep difﬁculties (trouble falling asleep, difﬁculty staying asleep, waking up too early, or waking up unrefreshed) 3 or more nights per week during the past month

Exclusion Criteria:

* Planned intervention (injection/ surgery/ new oral medications for pain or sleep) during the 4-week hBET use period
* Seizure disorder
* Photosensitivity
* Hearing or sight problems causing inability to use hBET
* Cognitive problems or dementia or mental health disorders causing inability to consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Qualitative semi-structured interviews | 5 weeks
  Interview at end of intervention period, following an interview guide, with responses thematically analysed

SECONDARY OUTCOMES:
Sleep and pain diary | 5 weeks
  Bespoke daily diary recording self reported pain and sleep
Actigraphy | 5 weeks
  Motion watch-based objective measure of gross sleep temporal parameters (total sleep time, sleep latency, wakenings after sleep onset, sleep efficiency)
Brief Pain Inventory | 5 weeks
  Gives two scores of 0-10 for pain severity and pain interference respectively, with 10 being worst in both cases.
Pittsburgh Sleep Quality Index | 5 weeks
  Gives a score of 0-21 with higher score indicating worse sleep quality
Hospital Anxiety and Depression Scale | 5 weeks
  Gives two scores of 0-21 for depression and anxiety respectively, with 21 being worst in both cases
Multidimensional Fatigue Inventory | 5 weeks
  Gives a score of 20-100, with higher scores indicating a higher level of fatigue
EuroQol 5 Dimensions (EQ-5D-5L) | 5 weeks
  A measure of global health state, providing a score of 1-5 in each of 5 domains (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), a global index score derived from population references ranging from 0-1 and a self reported description of overall health status on a 0-100 visual-analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halpin SJ, Casson AJ, Tang NKY, Jones AKP, O'Connor RJ, Sivan M. A feasibility study of pre-sleep audio and visual alpha brain entrainment for people with chronic pain and sleep disturbance. Front Pain Res (Lausanne). 2023 Feb 23;4:1096084. doi: 10.3389/fpain.2023.1096084. eCollection 2023. PMID 36910250